CLINICAL TRIAL: NCT00244764
Title: A Phase II Study of GW786034 Using a Randomised Discontinuation Design in Subjects With Locally Recurrent or Metastatic Clear-Cell Renal Cell Carcinoma
Brief Title: GW786034 In Subjects With Locally Recurrent Or Metastatic Clear Cell Renal Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VEG102616
Record Dates: First submitted 2005-10-25; First posted 2005-10-27 (Estimated); Results first posted 2011-01-25 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2015-09

CONDITIONS: Carcinoma, Renal Cell
Keywords: Angiogenesis; Renal Cell Carcinoma; Solid tumors; Pazopanib(GW786034)
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pazopanib (Experimental): All patients receive GW786034. At week 12, some subjects will be randomized based on response (SD) and the others will remain on drug. After the interim analysis, the design was changed to an open label, single arm study with all subjects receiving pazopanib.
  Interventions: Drug: GW786034
- Placebo (Placebo Comparator): All patients receive GW786034. At week 12, some subjects will be randomized based on response (SD) and the others will remain on drug. After the interim analysis, the design was changed to an open label, single arm study with all subjects receiving pazopanib.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GW786034 — All patients receive GW786034. At week 12, some subjects will be randomized based on response (SD) and the others will remain on drug. After the interim analysis, the design was changed to an open label, single arm study with all subjects receiving pazopanib.
  Arms: Pazopanib
Drug: Placebo — All patients receive GW786034. At week 12, some subjects will be randomized based on response (SD) and the others will remain on drug. After the interim analysis, the design was changed to an open label, single arm study with all subjects receiving pazopanib.
  Arms: Placebo

SUMMARY:
Phase II, multi-center, two-stage study utilising a randomised discontinuation design to evaluate the safety and efficacy of GW786034 (pazopanib) in adult subjects with locally recurrent or metastatic clear-cell Renal Cell Carcinoma (RCC). After the interim analysis, the design was changed to an open label, single arm study with all subjects receiving pazopanib.

ELIGIBILITY:
Inclusion criteria:

* Histologically or cytologically confirmed diagnosis of Renal Cell Carcinoma of predominantly clear-cell histology (excluding chromophobe, papillary, collecting duct, and undifferentiated tumors) which is metastatic or locally recurrent
* Either no prior systemic therapy or failed only 1 prior cytokine-based or bevacizumab-based therapy
* Evidence of documented measurable disease by RECIST criteria
* Male or female at least 21 years of age

A woman is eligible to enter and participate in the study if she is of:

1. Non-childbearing potential (i.e., physiologically incapable of becoming pregnant), including any female who:

   * Has had a hysterectomy,
   * Has had a bilateral oophorectomy (ovariectomy),
   * Has had a bilateral tubal ligation,
   * Is post-menopausal (total cessation of menses for >= 1 year).
2. Childbearing potential, has a negative serum pregnancy test at Screening Period and serum or urine pregnancy test at Day1, and agrees to use adequate contraception. GSK acceptable contraceptive methods, when used consistently and in accordance with both the product label and the instructions of the physician, are as follows:

   * An intrauterine device (IUD) with a documented failure rate of less than 1% per year.
   * Vasectomized partner who is sterile prior to the female subject's entry and is the sole sexual partner for that female.
   * Complete abstinence from sexual intercourse for 14 days before exposure to investigation product, through the clinical trial, and for at least 21 days after the last dose of investigational product.
   * Double-barrier contraception (condom with spermicidal jelly, foam suppository, or film; diaphragm with spermicide; or male condom and diaphragm with spermicide).

A man with a female partner of childbearing potential is eligible to enter and participate in the study if he uses a barrier method of contraception (e.g. condom) or abstinence during the study and for 28 days following the last dose of investigational drug.

* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0 or 1.
* Adequate bone marrow function.
* Adequate hepatic function.
* Adequate renal function.
* Adequate PT/PTT or INR/aPTT.
* Able to swallow and retain oral medications.
* Written informed consent.

Exclusion criteria:

* Received prior non-cytokine or non-bevacizumab therapies .
* Received chemotherapy for renal cell carcinoma.
* Have had any major surgery, radiotherapy, or immunotherapy within the last 28 days and/or not recovered from prior therapy.
* History of hypercalcemia within two months of start of therapy.
* Patients who are pregnant or lactating.
* Poorly controlled hypertension.
* QTc prolongation defined as a QTc interval ≥ 480 msecs or other significant ECG abnormalities.
* Has Class II, III or IV heart failure as defined by the New York Heart Association functional classification system. A subject who has a history of Class II heart failure and is asymptomatic on treatment may be considered eligible.
* Any history of cerebrovascular accident [CVA].
* History of myocardial infarction, admission for unstable angina, cardiac angioplasty or stenting within the last 12 weeks.
* History of venous thrombosis in last 12 weeks.
* Current use of therapeutic warfarin.
* Use of antiplatelet agents other than aspirin (≤ 325 mg/day).
* Leptomeningeal or brain metastases.
* Prior history of malignancies other than renal cell carcinoma (except for basal cell or squamous cell carcinoma of the skin, carcinoma in situ of the cervix or breast, or the subject has been free of any other malignancies for > 5 years).
* Any serious and/or unstable pre-existing medical, psychiatric, or other condition (including lab abnormalities) that could interfere with subject safety or obtaining informed consent.
* History of malabsorption syndrome, disease significantly affecting gastrointestinal function or major resection of the stomach or small bowel that could affect absorption, distribution, metabolism or excretion of study drugs. Has any unresolved bowel obstruction or diarrhea.
* Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol.
* Is on any specifically prohibited medication or requires any of these medications during treatment with GW786034.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2005-10; Primary Completion 2008-03 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (41):
- United States (11):
  - GSK Investigational Site, Duarte, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Orange, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Aurora, Colorado
  - GSK Investigational Site, Tucker, Georgia
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Dallas, Texas
- Australia (7):
  - GSK Investigational Site, Camperdown, New South Wales
  - GSK Investigational Site, Kogarah, New South Wales
  - GSK Investigational Site, Randwick, New South Wales
  - GSK Investigational Site, East Melbourne, Victoria
  - GSK Investigational Site, Footscay, Victoria
  - GSK Investigational Site, Heidelberg, Victoria
  - GSK Investigational Site, Parkville, Victoria
- Belgium (6):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Jette
  - GSK Investigational Site, Liège
  - GSK Investigational Site, Roeselare
  - GSK Investigational Site, Wilrijk
- China (6):
  - GSK Investigational Site, Guangzhou, Guangdong
  - GSK Investigational Site, Nanjing, Jiangsu
  - GSK Investigational Site, Jinan, Shandong
  - GSK Investigational Site, Hangzhou, Zhejiang
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Shanghai
- Czechia (3):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Hradec Králové
  - GSK Investigational Site, Prague
- Hong Kong (3):
  - GSK Investigational Site, Hong Kong
  - GSK Investigational Site, Kowloon
  - GSK Investigational Site, Tuenmen
- Israel (4):
  - GSK Investigational Site, Haifa
  - GSK Investigational Site, Petah Tikva
  - GSK Investigational Site, Tel Aviv
  - GSK Investigational Site, Zrifin
- GSK Investigational Site, Taipei, Taiwan

REFERENCES:
- [Background] Bonate PL, Suttle AB. Modeling tumor growth kinetics after treatment with pazopanib or placebo in patients with renal cell carcinoma. Cancer Chemother Pharmacol. 2013 Jul;72(1):231-40. doi: 10.1007/s00280-013-2191-0. Epub 2013 May 29. PMID 23715625
- [Background] Hutson TE, Davis ID, Machiels JP, De Souza PL, Rottey S, Hong BF, Epstein RJ, Baker KL, McCann L, Crofts T, Pandite L, Figlin RA. Efficacy and safety of pazopanib in patients with metastatic renal cell carcinoma. J Clin Oncol. 2010 Jan 20;28(3):475-80. doi: 10.1200/JCO.2008.21.6994. Epub 2009 Dec 14. PMID 20008644
- [Background] Tran HT, Liu Y, Zurita AJ, Lin Y, Baker-Neblett KL, Martin AM, Figlin RA, Hutson TE, Sternberg CN, Amado RG, Pandite LN, Heymach JV. Prognostic or predictive plasma cytokines and angiogenic factors for patients treated with pazopanib for metastatic renal-cell cancer: a retrospective analysis of phase 2 and phase 3 trials. Lancet Oncol. 2012 Aug;13(8):827-37. doi: 10.1016/S1470-2045(12)70241-3. Epub 2012 Jul 2. PMID 22759480
- [Background] White AJ, LaGerche A, Toner GC, Whitbourn RJ. Apical ballooning syndrome during treatment with a vascular endothelial growth factor receptor antagonist. Int J Cardiol. 2009 Jan 24;131(3):e92-4. doi: 10.1016/j.ijcard.2007.07.066. Epub 2007 Oct 24. PMID 17920711
- [Background] Xu CF, Reck BH, Goodman VL, Xue Z, Huang L, Barnes MR, Koshy B, Spraggs CF, Mooser VE, Cardon LR, Pandite LN. Association of the hemochromatosis gene with pazopanib-induced transaminase elevation in renal cell carcinoma. J Hepatol. 2011 Jun;54(6):1237-43. doi: 10.1016/j.jhep.2010.09.028. Epub 2011 Feb 12. PMID 21145803
- [Background] Xu CF, Reck BH, Xue Z, Huang L, Baker KL, Chen M, Chen EP, Ellens HE, Mooser VE, Cardon LR, Spraggs CF, Pandite L. Pazopanib-induced hyperbilirubinemia is associated with Gilbert's syndrome UGT1A1 polymorphism. Br J Cancer. 2010 Apr 27;102(9):1371-7. doi: 10.1038/sj.bjc.6605653. Epub 2010 Apr 13. PMID 20389299
- [Derived] Goldstein D, Rosenberg JE, Figlin RA, Townsend RR, McCann L, Carpenter C, Pandite L. Is change in blood pressure a biomarker of pazopanib and sunitinib efficacy in advanced/metastatic renal cell carcinoma? Eur J Cancer. 2016 Jan;53:96-104. doi: 10.1016/j.ejca.2015.10.006. Epub 2015 Dec 15. PMID 26702763

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was originally designed as a Phase II, multi-centre study utilizing a randomized discontinuation design. In the original study design, a 12-week Lead-in Phase was an open-label period during which all enrolled participans received pazopanib.
Pre-assignment Details: All participants began with 12 weeks of open-label treatment. In the original design, participants with stable disease at Week 12 were to be randomized. After the interim analysis, the study was amended to be treated like a single-arm open-label study. Any participants who had been randomized to placebo were to be crossed back to pazopanib.
Groups:
- Pazopanib 800 mg: Pazopanib 800 milligrams (mg) (tablets) administered orally once a day
Period: Overall Study
Arm/Group | Pazopanib 800 mg
Started | 225
Completed | 129
Not Completed | 96
Not completed — Adverse Event | 37
Not completed — Lost to Follow-up | 23
Not completed — Withdrawal by Subject | 12
Not completed — Disease Progression | 13
Not completed — Protocol Violation | 2
Not completed — Death | 1
Not completed — Off Study Medication for >21 Days | 1
Not completed — Declining Performance Status | 1
Not completed — Participant was Hospitalized until Death | 1
Not completed — Primary Investigator Discretion | 2
Not completed — Sponsor Terminated Study | 2
Not completed — Developed Secondary Malignancy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pazopanib 800 mg
Number analyzed (Participants) | 225
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.8 (10.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69
  Male | 156
Race/Ethnicity, Customized [Number; unit: participants]
  White | 178
  Asian-Japanese/East Asian/South East Asian HER | 38
  African American/African Heritage (HER) | 4
  Asian-Central/South Asian Heritage | 2
  American Indian or Alaska Native and White | 1
  Asian-Mixed Asian Heritage | 1
  Native Hawaiian or other Pacific Islander | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Response by RECIST Criteria
Description: The overall response is the number of participants who experience a confirmed complete (CR) or partial response (PR) of the total analysis population. Per the Response Evaluation Criteria In Solid Tumors (RECIST): CR = all detectable tumor has disappeared, PR = a >=30% decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum, Progressive disease (PD) = a >=20% increase in target lesions, Stable Disease = small changes that do not meet previously given criteria.
Time Frame: Baseline to Response (up to 2.40 years). Assessments occurred at Week 12 and every 8 weeks thereafter.
Population: All Enrolled: all participants who received at least one dose of pazopanib
Measure: Number; unit: participants
Arm/Group | Pazopanib 800 mg
Number analyzed (Participants) | 225
participants
  Complete Response | 3
  Partial Response | 75
  Stable Disease | 101
  Progressive Disease | 24
  Not evaluable | 22
  Complete Response + Partial Response | 78
Statistical Analysis 1: Comparison: Pazopanib 800 mg; Test type: Superiority or Other; percentage = 34.7, 95% CI [28.4 to 40.9] — The estimated value provided is the response rate

2. Primary Outcome: Stable Disease at 12 Weeks - Interim Analysis of First 60 Participants
Description: The protocol called for an interim analysis of the first 60 participants to determine their status at Week 12, and to determine the number of participants with stable disease, although all categories were reported. Stable disease is defined as a disease that has not grown enough to be called progressive disease and has not shrunk enough to be called partial/complete response.
Time Frame: Week 12
Population: Subset of the All Enrolled Population including only the first 60 participants
Measure: Number; unit: participants
Arm/Group | Pazopanib 800 mg
Number analyzed (Participants) | 60
participants
  Complete Response | 0
  Partial Response | 23
  Stable Disease | 25
  Progressive Disease | 3
  Unknown | 9
Statistical Analysis 1: Comparison: Pazopanib 800 mg; Test type: Superiority or Other; percentage = 42, 95% CI [29 to 54] — The estimated value is the percentage of the first 60 participants who had stable disease at Week 12, as assessed by the investigator

3. Secondary Outcome: Duration of Response
Description: Using RECIST criteria: date of first confirmed tumor response (CR or PR) to date of tumor progression or to death. Participants who did not progress or die were censored at their last radiologic assessment. Only participants who had a response were analyzed.
Time Frame: First response until progression of disease (up to 2.40 years). Assessments occurred at Week 12 and every 8 weeks thereafter.
Population: All participants in the Enrolled Population who had a CR or PR
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Pazopanib 800 mg
Number analyzed (Participants) | 78
weeks | 68 [53.7 to NA] — There were too few responses with a known end date to calculate the upper bound of the 95% confidence interval.

4. Secondary Outcome: Progression-free Survival
Description: Progression-free Survival is defined as the interval between the first day of treatment and the earliest date of disease progression or death due to any cause, whichever occurred first. Progressive disease is defined as a >=20% increase in target lesions.
Time Frame: From the first day of treatment to the earliest date of disease progression or death due to any cause (up to 2.40 years)
Population: All Enrolled Population. Participants who did not progress or die were censored at their last radiologic assessment.
Measure: Median (95% Confidence Interval); unit: weeks
Groups:
- Pazopanib 800 mg: Pazopanib 800 mg (tablets) administered orally once a day
Arm/Group | Pazopanib 800 mg
Number analyzed (Participants) | 225
weeks | 45.3 [36.0 to 59.1]

ADVERSE EVENTS:
Time Frame: Until participant was off study, approximately 7.84 years
Arm/Group | Pazopanib 800 mg
Serious Adverse Events (participants affected / at risk) | 80/225
Other Adverse Events (participants affected / at risk) | 215/225
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pazopanib 800 mg (N=225)
Abdominal pain (Gastrointestinal disorders) | 3
Diarrhhoea (Gastrointestinal disorders) | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3
Large intestine perforation (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Abdominal pain lower (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Faecaloma (Gastrointestinal disorders) | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1
Ileal perforation (Gastrointestinal disorders) | 1
Oesophagitis (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 3
Hyponatraemia (Metabolism and nutrition disorders) | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Chest pain (General disorders) | 4
Fatigue (General disorders) | 2
General physical health deterioration (General disorders) | 1
Oedema peripheral (General disorders) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Post procedural complication (Injury, poisoning and procedural complications) | 1
Postoperative wound complication (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 2
Cerebrovascular accident (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Haemorrhage intracranial (Nervous system disorders) | 1
Nerve root compression (Nervous system disorders) | 1
Alanine aminotransferase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 2
Body temperature increased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Lipase increased (Investigations) | 3
Anal abscess (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Atrial fibrillation (Cardiac disorders) | 2
Myocardial infarction (Cardiac disorders) | 2
Stress cardiomyopathy (Cardiac disorders) | 1
Ventricular fibrillation (Cardiac disorders) | 1
Bile duct stenosis (Hepatobiliary disorders) | 1
Bile duct stone (Hepatobiliary disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1
Jaundice (Hepatobiliary disorders) | 1
Hypertension (Vascular disorders) | 2
Deep vein thrombosis (Vascular disorders) | 1
Haematoma (Vascular disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Haemangioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Confusional state (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Hydrocele (Congenital, familial and genetic disorders) | 1
Retinal tear (Eye disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Large intestinal stenosis (Gastrointestinal disorders) | 1
Large intestinal ulcer (Gastrointestinal disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Stab wound (Injury, poisoning and procedural complications) | 1
Headache (Nervous system disorders) | 1
Blood creatinine increased (Investigations) | 1
Blood thyroid stimulating hormone decreased (Investigations) | 1
Blood urea increased (Investigations) | 1
Ejection fraction decreased (Investigations) | 1
Cellulitis (Infections and infestations) | 1
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Haematuria (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Pelvic pain (Reproductive system and breast disorders) | 1
Urogenital haemorrhage (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pazopanib 800 mg (N=225)
Diarrhoea (Gastrointestinal disorders) | 148
Nausea (Gastrointestinal disorders) | 99
Vomiting (Gastrointestinal disorders) | 50
Abdominal pain (Gastrointestinal disorders) | 37
Constipation (Gastrointestinal disorders) | 37
Dyspepsia (Gastrointestinal disorders) | 25
Flatulence (Gastrointestinal disorders) | 14
Hair colour changes (Skin and subcutaneous tissue disorders) | 100
Rash (Skin and subcutaneous tissue disorders) | 37
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 25
Alopecia (Skin and subcutaneous tissue disorders) | 26
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 14
Dry skin (Skin and subcutaneous tissue disorders) | 14
Erythema (Skin and subcutaneous tissue disorders) | 12
Fatigue (General disorders) | 108
Oedema peripheral (General disorders) | 20
Dysgeusia (Nervous system disorders) | 57
Headache (Nervous system disorders) | 47
Dizziness (Nervous system disorders) | 31
Hypertension (Vascular disorders) | 99
Cough (Respiratory, thoracic and mediastinal disorders) | 44
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 26
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 25
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 12
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 15
Arthralgia (Musculoskeletal and connective tissue disorders) | 35
Back pain (Musculoskeletal and connective tissue disorders) | 28
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 12
Muscle spasms (Musculoskeletal and connective tissue disorders) | 19
Pain in extremity (Musculoskeletal and connective tissue disorders) | 20
Myalgia (Musculoskeletal and connective tissue disorders) | 12
Decreased appetite (Metabolism and nutrition disorders) | 69
Upper respiratory tract infection (Infections and infestations) | 22
Nasopharyngitis (Infections and infestations) | 18
Alanine aminotransferase increased (Investigations) | 32
Aspartate aminotransferase increased (Investigations) | 28
Weight decreased (Investigations) | 23
Insomnia (Psychiatric disorders) | 21
Anxiety (Psychiatric disorders) | 13
Anaemia (Blood and lymphatic system disorders) | 12
Abdominal pain upper (Gastrointestinal disorders) | 13
Stomatitis (Gastrointestinal disorders) | 13
Abdominal distension (Gastrointestinal disorders) | 12
Chest pain (General disorders) | 16
Pyrexia (General disorders) | 16
Asthenia (General disorders) | 14
Mucosal inflammation (General disorders) | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.